CLINICAL TRIAL: NCT00294047
Title: A Study to Evaluate Safety, Immunogenicity and Efficacy of GSK Biologicals HPV-16/18 L1/AS04 Vaccine Administered Intramuscularly According to a Three-dose Schedule (0, 1, 6 Month) in Healthy Adult Female Subjects Aged 26 Years and Above
Brief Title: Study to Evaluate the Efficacy of the Human Papillomavirus Vaccine in Healthy Adult Women of 26 Years of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 104820; 2005-002546-20 (EudraCT Number)
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Results first posted 2012-03-27 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Infections, Papillomavirus; Papillomavirus Vaccines
Keywords: Vaccine; Human papillomavirus; Cervical Cancer; Cervical Infection
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Cervarix Group (Experimental): Subjects received 3 doses of Cervarix™ vaccine. Cervarix vaccine was administered intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6 months schedule.
  Interventions: Biological: Cervarix
- Aluminium Hydroxide Group (Placebo Comparator): Subjects received 3 doses of Aluminium Hydroxide [Al(OH)3]. Aluminium Hydroxide was administered intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6 months schedule.
  Interventions: Biological: Placebo control

INTERVENTIONS:
Biological: Cervarix — Subjects were planned to receive three doses of the study vaccine administered intramuscularly according to a 0, 1, 6 month vaccination schedule.
  Arms: Cervarix Group
Biological: Placebo control — Subjects were planned to receive three doses of the control vaccine administered intramuscularly according to a 0, 1, 6 month vaccination schedule.
  Arms: Aluminium Hydroxide Group

SUMMARY:
This is a multicentre study in which women were planned to receive either the Human Papillomavirus Vaccine (HPV) vaccine or control. Under Protocol Amendment 3, study participation will last approximately 48 months and involves a total of eleven scheduled visits. Under Protocol Amendment 4, study participation will last up to 84 months and involves a maximum of seventeen scheduled visits.

DETAILED DESCRIPTION:
The Protocol Posting has been updated due to protocol amendment 5 and in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion criteria:

* A woman who the investigator believes that she can and will comply with the requirements of the protocol.
* A women of at least 26 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to enrolment.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Subject must have intact cervix.
* Subject must have a negative urine pregnancy test. This test is not applicable to women of non-childbearing potential.
* Subject must be of non-childbearing potential or, if of childbearing potential, she must be abstinent or must be using an effective method of birth control for 30 days prior to the first vaccination and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion criteria:

* Pregnant or breastfeeding (women must be at least three months post-pregnancy and not breastfeeding to enter the study).
* A women planning to become pregnant, likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive precautions during the vaccination phase of the study, i.e. up to two months after the last vaccine dose (Month 0 - 8).
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period (up to Month 84).
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after (i.e. days 0 - 29) the first dose of study vaccine. Planned administration/administration of routine vaccines up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Previous administration of components of the investigational vaccine
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* History of HPV infection/treatment or planned treatment to evaluate an abnormal cervical cytology (Pap smear) test, e.g. colposcopy.
* Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccine.
* Hypersensitivity to latex.
* Known acute or chronic, clinically significant neurologic, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* History of chronic condition(s) requiring treatment.
* Administration of immunoglobulins and/or any blood product within three months preceding the first dose of study vaccine, or planned administration during the study period. Enrolment will be deferred until the subject is outside of specified window.
* Acute disease at the time of enrolment.
* Heavy bleeding (menstruation or other) or heavy vaginal discharge in which a pelvic exam cannot be performed (and no cervical sample can be taken). Enrolment will be deferred until condition is resolved according to investigators medical judgement.

Min Age: 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5752 (Actual)
Dates: Start 2006-02-16 (Actual); Primary Completion 2014-01-29 (Actual); Study Completion 2014-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (66):
- United States (32):
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, New Bern, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Wexford, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, Wenatchee, Washington
  - GSK Investigational Site, La Crosse, Wisconsin
- Australia (2):
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Perth, Western Australia
- Canada (7):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Mexico (2):
  - GSK Investigational Site, Cuenavaca, Morelos
  - GSK Investigational Site, Jojutla / Morelos
- Netherlands (3):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Delft
  - GSK Investigational Site, Rotterdam
- GSK Investigational Site, Lima, Peru
- Philippines (3):
  - GSK Investigational Site, Laguna
  - GSK Investigational Site, San Pablo
  - GSK Investigational Site, Taft Avenue, Manila
- Portugal (5):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
  - GSK Investigational Site, Setúbal
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yekaterinburg
- GSK Investigational Site, Singapore, Singapore
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (6):
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Gateshead
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=1517

REFERENCES:
- [Background] Descamps D, Hardt K, Spiessens B, Izurieta P, Verstraeten T, Breuer T, Dubin G. Safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine for cervical cancer prevention: a pooled analysis of 11 clinical trials. Hum Vaccin. 2009 May;5(5):332-40. doi: 10.4161/hv.5.5.7211. Epub 2009 May 20. PMID 19221517
- [Background] Skinner SR, Szarewski A, Romanowski B, Garland SM, Lazcano-Ponce E, Salmeron J, Del Rosario-Raymundo MR, Verheijen RH, Quek SC, da Silva DP, Kitchener H, Fong KL, Bouchard C, Money DM, Ilancheran A, Cruickshank ME, Levin MJ, Chatterjee A, Stapleton JT, Martens M, Quint W, David MP, Meric D, Hardt K, Descamps D, Geeraerts B, Struyf F, Dubin G; VIVIANE Study Group. Efficacy, safety, and immunogenicity of the human papillomavirus 16/18 AS04-adjuvanted vaccine in women older than 25 years: 4-year interim follow-up of the phase 3, double-blind, randomised controlled VIVIANE study. Lancet. 2014 Dec 20;384(9961):2213-27. doi: 10.1016/S0140-6736(14)60920-X. Epub 2014 Sep 1. PMID 25189358
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- [Background] Wheeler CM, Skinner SR, Del Rosario-Raymundo MR, Garland SM, Chatterjee A, Lazcano-Ponce E, Salmeron J, McNeil S, Stapleton JT, Bouchard C, Martens MG, Money DM, Quek SC, Romanowski B, Vallejos CS, Ter Harmsel B, Prilepskaya V, Fong KL, Kitchener H, Minkina G, Lim YKT, Stoney T, Chakhtoura N, Cruickshank ME, Savicheva A, da Silva DP, Ferguson M, Molijn AC, Quint WGV, Hardt K, Descamps D, Suryakiran PV, Karkada N, Geeraerts B, Dubin G, Struyf F; VIVIANE Study Group. Efficacy, safety, and immunogenicity of the human papillomavirus 16/18 AS04-adjuvanted vaccine in women older than 25 years: 7-year follow-up of the phase 3, double-blind, randomised controlled VIVIANE study. Lancet Infect Dis. 2016 Oct;16(10):1154-1168. doi: 10.1016/S1473-3099(16)30120-7. Epub 2016 Jun 28. PMID 27373900
- [Background] Wheeler CM, Struyf F; HPV-015 study group. The safety of Cervarix? - Authors' reply. Lancet Infect Dis. 2017 Jan;17(1):20-21. doi: 10.1016/S1473-3099(16)30540-0. No abstract available. PMID 27998562
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Chen J, Gopala K, Akarsh PK, Struyf F, Rosillon D. Prevalence and Incidence of Human Papillomavirus (HPV) Infection Before and After Pregnancy: Pooled Analysis of the Control Arms of Efficacy Trials of HPV-16/18 AS04-Adjuvanted Vaccine. Open Forum Infect Dis. 2019 Dec 4;6(12):ofz486. doi: 10.1093/ofid/ofz486. eCollection 2019 Dec. PMID 31824976
- [Derived] Rosillon D, Baril L, Del Rosario-Raymundo MR, Wheeler CM, Skinner SR, Garland SM, Salmeron J, Lazcano-Ponce E, Vallejos CS, Stoney T, Ter Harmsel B, Lim TYK, Quek SC, Minkina G, McNeil SA, Bouchard C, Fong KL, Money D, Ilancheran A, Savicheva A, Cruickshank M, Chatterjee A, Fiander A, Martens M, Bozonnat MC, Struyf F, Dubin G, Castellsague X. Risk of newly detected infections and cervical abnormalities in adult women seropositive or seronegative for naturally acquired HPV-16/18 antibodies. Cancer Med. 2019 Aug;8(10):4938-4953. doi: 10.1002/cam4.1879. Epub 2019 Jul 5. PMID 31273942
- [Derived] Skinner SR, Wheeler CM, Romanowski B, Castellsague X, Lazcano-Ponce E, Del Rosario-Raymundo MR, Vallejos C, Minkina G, Pereira Da Silva D, McNeil S, Prilepskaya V, Gogotadze I, Money D, Garland SM, Romanenko V, Harper DM, Levin MJ, Chatterjee A, Geeraerts B, Struyf F, Dubin G, Bozonnat MC, Rosillon D, Baril L; VIVIANE Study Group. Progression of HPV infection to detectable cervical lesions or clearance in adult women: Analysis of the control arm of the VIVIANE study. Int J Cancer. 2016 May 15;138(10):2428-38. doi: 10.1002/ijc.29971. PMID 26685704
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Some subjects completed the study at Months 36 and 48 as they did not want to participate to the extensions up to Month 84, but they were included in the safety analysis for these subsequent timepoints.
Pre-assignment Details: Enrolment was stratified by (1) age, with the majority of subjects in age strata 26 - 35 years and 36 - 45 years (about 45% each) and about 10% in the age stratum 46+ years, and (2) previous HPV history (in each age stratum, the number of women with a history of HPV infection/treatment was limited to approximately 15%).
Period: Month 48
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Started | 2881 | 2871
Participated up to Month 48 | 2305 | 2281
Completed | 2456 | 2438
Not Completed | 425 | 433
Not completed — Adverse Event | 28 | 13
Not completed — Protocol Violation | 4 | 4
Not completed — Withdrawal by Subject | 111 | 115
Not completed — Lost to Follow-up | 272 | 287
Not completed — Other | 10 | 14
Period: Month 84
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Started | 2877 | 2870
Completed | 1904 (The number of subjects who remained up to Month 48 in the Cervarix Group = 2146) | 1881 (The number of subjects who remained up to Month 48 in the Aluminium Hydroxide Group = 2116)
Not Completed | 973 | 989
Not completed — Adverse Event | 4 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 33 | 31
Not completed — Lost to Follow-up | 187 | 190
Not completed — Absent Cervix | 2 | 0
Not completed — Work related reasons | 4 | 2
Not completed — Center closed, subject did not transfer | 1 | 0
Not completed — Family problems | 2 | 2
Not completed — Lack of time | 3 | 1
Not completed — Personal reason | 2 | 4
Not completed — Subject does not want male physician | 1 | 0
Not completed — Transport reimbursement delayed | 0 | 1
Not completed — Unable to reach study site | 1 | 0
Not completed — Under investigation locally | 1 | 0
Not completed — Visit missed | 0 | 1
Not completed — No consent for Month 84 Follow-up | 731 | 754

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Aluminium Hydroxide Group | Total
Number analyzed (Participants) | 2881 | 2871 | 5752
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.0 (7.24) | 37.0 (7.32) | 37.0 (7.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2881 | 2871 | 5752
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Human Papillomavirus (HPV)-16 or HPV-18 and/or With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 and/or -18 Cervical Infection.
Description: CIN1+ = CIN grades 1, 2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Persistent HPV infection = detection of the same HPV type(s) by polymerase chain reaction (PCR) in cervical samples at 2 consecutive evaluations over approximately a 6-month interval.
  * DNA- and sero-/+: subjects HPV deoxyribonucleic acid (DNA) negative (DNA-) at Month 0 and 6 and seronegative/positive (sero-/+) at Month 0 for the corresponding HPV-type by Enzyme-linked Immunosorbent Assay (ELISA)
  * Overall: subjects DNA- at Month 0 and 6 for the corresponding HPV-type, regardless of initial serostatus
Time Frame: Up to Month 48
Population: The According-To-Protocol cohort for efficacy included subjects who had a normal or low-grade cytology (negative or atypical squamous cells of undetermined significance (ASC-US) or low-grade squamous intraepithelial lesion (LSIL)) at Month 0, who received 3 doses. A 15% subset of women enrolled with prior history of HPV infection was excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2224 | 2190
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1898 | 1854
  HPV-16/18, DNA- and sero- subjects | 7 | 36
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1545 | 1521
  HPV-16, DNA- and sero- subjects | 5 | 27
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1597 | 1571
  HPV-18, DNA- and sero- subjects | 2 | 10
  HPV-16/18, DNA- and sero+ subjects: number analyzed (Participants) | 900 | 864
  HPV-16/18, DNA- and sero+ subjects | 2 | 14
  HPV-16, DNA- and sero+ subjects: number analyzed (Participants) | 605 | 594
  HPV-16, DNA- and sero+ subjects | 1 | 9
  HPV-18, DNA- and sero+ subjects: number analyzed (Participants) | 574 | 550
  HPV-18, DNA- and sero+ subjects | 1 | 5
  HPV-16/18, overall | 9 | 51
  HPV-16, overall: number analyzed (Participants) | 2167 | 2131
  HPV-16, overall | 6 | 36
  HPV-18, overall: number analyzed (Participants) | 2203 | 2165
  HPV-18, overall | 3 | 16

2. Primary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With HPV-16 or HPV-18 and/or With Histopathologically-CIN1+ Associated With HPV-16 and/or -18 Cervical Infection Detected Using the HPV Type Assignment Algorithm (TAA).
Description: CIN1+ = CIN grades 1, 2 and 3, AIS and invasive cervical cancer. Persistent cervical HPV infection (6-month definition) = detection of the same HPV type(s) by PCR in cervical samples at 2 consecutive evaluations over approximately a 6-month interval.
  * DNA- and sero-/+: subjects HPV DNA negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative/positive (sero-/+) for HPV-16 and/or HPV-18 by ELISA at baseline (Month 0).
  * Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
Time Frame: Up to Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2224 | 2190
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1898 | 1854
  HPV-16/18, DNA- and sero- subjects | 7 | 36
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1545 | 1521
  HPV-16, DNA- and sero- subjects | 5 | 27
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1597 | 1571
  HPV-18, DNA- and sero- subjects | 2 | 10
  HPV-16/18, DNA- and sero+ subjects: number analyzed (Participants) | 900 | 864
  HPV-16/18, DNA- and sero+ subjects | 2 | 12
  HPV-16, DNA- and sero+ subjects: number analyzed (Participants) | 605 | 594
  HPV-16, DNA- and sero+ subjects | 1 | 8
  HPV-18, DNA- and sero+ subjects: number analyzed (Participants) | 574 | 550
  HPV-18, DNA- and sero+ subjects | 1 | 4
  HPV-16/18, overall | 9 | 49
  HPV-16, overall: number analyzed (Participants) | 2167 | 2131
  HPV-16, overall | 6 | 35
  HPV-18, overall: number analyzed (Participants) | 2203 | 2165
  HPV-18, overall | 3 | 15

3. Primary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Human Papillomavirus (HPV)-16 or HPV-18 and/or With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 and/or -18 Cervical Infection.
Description: CIN1+ = CIN grades 1, 2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer. Persistent HPV infection = detection of the same HPV type(s) by polymerase chain reaction (PCR) in cervical samples at 2 consecutive evaluations over approximately a 6-month interval. - DNA- and sero-/+: subjects HPV deoxyribonucleic acid (DNA) negative (DNA-) at Month 0 and 6 and seronegative/positive (sero-/+) at Month 0 for the corresponding HPV-type by Enzyme-linked Immunosorbent Assay (ELISA) - Overall: subjects DNA- at Month 0 and 6 for the corresponding HPV-type, regardless of initial serostatus
Time Frame: Up to Month 84
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2168 | 2147
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1852 | 1818
  HPV-16/18, DNA- and sero- subjects | 7 | 71
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1507 | 1491
  HPV-16, DNA- and sero- subjects | 5 | 53
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1565 | 1541
  HPV-18, DNA- and sero- subjects | 3 | 20
  HPV-16/18, DNA- and sero+ subjects: number analyzed (Participants) | 870 | 849
  HPV-16/18, DNA- and sero+ subjects | 3 | 16
  HPV-16, DNA- and sero+ subjects: number analyzed (Participants) | 588 | 584
  HPV-16, DNA- and sero+ subjects | 2 | 10
  HPV-18, DNA- and sero+ subjects: number analyzed (Participants) | 552 | 540
  HPV-18, DNA- and sero+ subjects | 1 | 6
  HPV-16/18, overall | 10 | 90
  HPV-16, overall: number analyzed (Participants) | 2112 | 2091
  HPV-16, overall | 7 | 63
  HPV-18, overall: number analyzed (Participants) | 2149 | 2123
  HPV-18, overall | 4 | 29

4. Primary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With HPV-16 or HPV-18 and/or With Histopathologically-CIN1+ Associated With HPV-16 and/or -18 Cervical Infection Detected Using the HPV Type Assignment Algorithm (TAA).
Description: CIN1+ = CIN grades 1, 2 and 3, AIS and invasive cervical cancer. Persistent cervical HPV infection (6-month definition) = detection of the same HPV type(s) by PCR in cervical samples at 2 consecutive evaluations over approximately a 6-month interval. - DNA- and sero-/+: subjects HPV DNA negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative/positive (sero-/+) for HPV-16 and/or HPV-18 by ELISA at baseline (Month 0). - Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
Time Frame: Up to Month 84
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2168 | 2147
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1852 | 1818
  HPV-16/18, DNA- and sero- subjects | 7 | 71
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1507 | 1491
  HPV-16, DNA- and sero- subjects | 5 | 53
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1565 | 1541
  HPV-18, DNA- and sero- subjects | 2 | 20
  HPV-16/18, DNA- and sero+ subjects: number analyzed (Participants) | 870 | 849
  HPV-16/18, DNA- and sero+ subjects | 3 | 14
  HPV-16, DNA- and sero+ subjects: number analyzed (Participants) | 588 | 584
  HPV-16, DNA- and sero+ subjects | 2 | 9
  HPV-18, DNA- and sero+ subjects: number analyzed (Participants) | 552 | 540
  HPV-18, DNA- and sero+ subjects | 1 | 5
  HPV-16/18, overall | 10 | 88
  HPV-16, overall: number analyzed (Participants) | 2112 | 2091
  HPV-16, overall | 7 | 62
  HPV-18, overall: number analyzed (Participants) | 2149 | 2123
  HPV-18, overall | 3 | 28

5. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Human Papillomavirus (HPV)-16 or HPV-18
Description: Persistent cervical HPV infection (6-month definition) was defined as the detection of the same HPV type(s) by PCR in cervical samples at 2 consecutive evaluations over approximately a 6-month interval.
  Detection was done in:
  * DNA- and sero-/+: subjects HPV DNA negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative/positive (sero-/+) for HPV-16 and/or HPV-18 by ELISA at baseline (Month 0).
  * Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
Time Frame: Up to Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2178 | 2152
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1859 | 1822
  HPV-16/18, DNA- and sero- subjects | 6 | 34
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1518 | 1495
  HPV-16, DNA- and sero- subjects | 5 | 26
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1566 | 1542
  HPV-18, DNA- and sero- subjects | 1 | 8
  HPV-16/18, DNA- and sero+ subjects: number analyzed (Participants) | 880 | 851
  HPV-16/18, DNA- and sero+ subjects | 2 | 11
  HPV-16, DNA- and sero+ subjects: number analyzed (Participants) | 591 | 583
  HPV-16, DNA- and sero+ subjects | 1 | 8
  HPV-18, DNA- and sero+ subjects: number analyzed (Participants) | 562 | 543
  HPV-18, DNA- and sero+ subjects | 1 | 3
  HPV-16/18, overall | 8 | 45
  HPV-16, overall: number analyzed (Participants) | 2126 | 2094
  HPV-16, overall | 6 | 34
  HPV-18, overall: number analyzed (Participants) | 2160 | 2127
  HPV-18, overall | 2 | 11

6. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With Human Papillomavirus (HPV)-16 or HPV-18
Description: Persistent cervical HPV infection (12-month definition) was defined as the detection of the same HPV type(s) PCR in cervical samples at all available time points over approximately a 12-month interval (evaluations are planned at approximately 6-month intervals).
  * DNA- and sero-/+: subjects HPV DNA negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative/positive (sero-/+) for HPV-16 and/or HPV-18 by ELISA at baseline (Month 0).
  * Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
Time Frame: Up to Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2146 | 2124
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1832 | 1800
  HPV-16/18, DNA- and sero- subjects | 2 | 18
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1499 | 1476
  HPV-16, DNA- and sero- subjects | 1 | 12
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1543 | 1525
  HPV-18, DNA- and sero- subjects | 1 | 6
  HPV-16/18, DNA- and sero+ subjects: number analyzed (Participants) | 864 | 839
  HPV-16/18, DNA- and sero+ subjects | 0 | 3
  HPV-16, DNA- and sero+ subjects: number analyzed (Participants) | 579 | 577
  HPV-16, DNA- and sero+ subjects | 0 | 2
  HPV-18, DNA- and sero+ subjects: number analyzed (Participants) | 553 | 532
  HPV-18, DNA- and sero+ subjects | 0 | 1
  HPV-16/18, overall | 2 | 21
  HPV-16, overall: number analyzed (Participants) | 2095 | 2069
  HPV-16, overall | 1 | 14
  HPV-18, overall: number analyzed (Participants) | 2128 | 2099
  HPV-18, overall | 1 | 7

7. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Oncogenic HPV Types Individually or in Combinations.
Description: Persistent cervical HPV infection (6-month definition) = detection of the same HPV type(s) by PCR in cervical samples at 2 consecutive evaluations over approximately a 6-month interval.
  Oncogenic HPV types included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Detection was done in subjects HPV DNA- for the corresponding HPV type at baseline (at month 0 and Month 6) regardless of initial serostatus.
  HPV-HRW=All high-risk (oncogenic) HPV types excluding HPV-16 and HPV-18. HPV-HR=High-risk (oncogenic) HPV types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
Time Frame: Up to Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2179 | 2154
Participants
  HPV-16: number analyzed (Participants) | 2126 | 2094
  HPV-16 | 6 | 34
  HPV-18: number analyzed (Participants) | 2160 | 2127
  HPV-18 | 2 | 11
  HPV-31: number analyzed (Participants) | 2126 | 2132
  HPV-31 | 4 | 19
  HPV-33: number analyzed (Participants) | 2158 | 2136
  HPV-33 | 8 | 6
  HPV-35: number analyzed (Participants) | 2165 | 2144
  HPV-35 | 8 | 13
  HPV-39: number analyzed (Participants) | 2150 | 2119
  HPV-39 | 20 | 11
  HPV-45: number analyzed (Participants) | 2160 | 2130
  HPV-45 | 4 | 17
  HPV-51: number analyzed (Participants) | 2125 | 2113
  HPV-51 | 27 | 26
  HPV-52: number analyzed (Participants) | 2113 | 2101
  HPV-52 | 33 | 38
  HPV-56: number analyzed (Participants) | 2154 | 2123
  HPV-56 | 16 | 20
  HPV-58: number analyzed (Participants) | 2152 | 2135
  HPV-58 | 12 | 8
  HPV-59: number analyzed (Participants) | 2158 | 2126
  HPV-59 | 12 | 11
  HPV-66: number analyzed (Participants) | 2141 | 2122
  HPV-66 | 27 | 27
  HPV-68: number analyzed (Participants) | 2138 | 2128
  HPV-68 | 15 | 23
  HPV-31/45: number analyzed (Participants) | 2175 | 2152
  HPV-31/45 | 8 | 35
  HPV-31/45/33/52/58 | 58 | 83
  HPV-39/45/59/68 | 50 | 60
  HPV-31/33/35/52/58 | 63 | 80
  HPV-31/45/33/52/58/35/39/51/56/59 | 132 | 146
  HPV-HRW | 163 | 185
  HPV-HR | 170 | 217

8. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With Oncogenic HPV Types Individually or in Combinations.
Description: Persistent HPV infection (12-month definition) = detection of the same HPV type(s) by PCR in cervical samples at available time points over approximately a 12-month interval (evaluations are planned at approximately 6-month intervals).
  Oncogenic HPV types included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  subjects HPV DNA- for the corresponding HPV type at Month 0 6, regardless of initial serostatus.
  HPV-HRW=All high-risk (oncogenic) HPV types excluding HPV-16 and HPV-18 HPV-HR=High-risk (oncogenic) HPV types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 , 68
Time Frame: Up to Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2147 | 2126
Participants
  HPV-16: number analyzed (Participants) | 2095 | 2069
  HPV-16 | 1 | 14
  HPV-18: number analyzed (Participants) | 2128 | 2099
  HPV-18 | 1 | 7
  HPV-31: number analyzed (Participants) | 2096 | 2104
  HPV-31 | 2 | 10
  HPV-33: number analyzed (Participants) | 2126 | 2110
  HPV-33 | 5 | 5
  HPV-35: number analyzed (Participants) | 2133 | 2116
  HPV-35 | 3 | 8
  HPV-39: number analyzed (Participants) | 2119 | 2091
  HPV-39 | 12 | 5
  HPV-45: number analyzed (Participants) | 2129 | 2102
  HPV-45 | 4 | 8
  HPV-51: number analyzed (Participants) | 2093 | 2086
  HPV-51 | 11 | 14
  HPV-52: number analyzed (Participants) | 2081 | 2074
  HPV-52 | 21 | 23
  HPV-56: number analyzed (Participants) | 2124 | 2096
  HPV-56 | 4 | 8
  HPV-58: number analyzed (Participants) | 2120 | 2108
  HPV-58 | 8 | 7
  HPV-59: number analyzed (Participants) | 2126 | 2098
  HPV-59 | 4 | 3
  HPV-66: number analyzed (Participants) | 2109 | 2094
  HPV-66 | 10 | 8
  HPV-68: number analyzed (Participants) | 2106 | 2100
  HPV-68 | 7 | 13
  HPV-31/45: number analyzed (Participants) | 2144 | 2124
  HPV-31/45 | 6 | 17
  HPV-31/45/33/52/58 | 39 | 49
  HPV-39/45/59/68 | 27 | 29
  HPV-31/33/35/52/58 | 38 | 51
  HPV-31/45/33/52/58/35/39/51/56/59 | 70 | 84
  HPV-HRW | 86 | 105
  HPV-HR | 88 | 122

9. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)2+ Associated With HPV-16 and/or -18 Cervical Infection Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN2+ was defined as CIN grades 2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Detection was done in:
  * DNA- and sero-: subjects HPV deoxyribonucleic acid (DNA) negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative (sero-) for HPV-16 and/or HPV-18 by Enzyme-linked Immunosorbent Assay (ELISA) at baseline (Month 0).
  * Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
  Note: Results for seropositive status were not analysed.
Time Frame: Up to Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2224 | 2190
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1898 | 1854
  HPV-16/18, DNA- and sero- subjects | 0 | 4
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1545 | 1521
  HPV-16, DNA- and sero- subjects | 0 | 3
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1597 | 1571
  HPV-18, DNA- and sero- subjects | 0 | 2
  HPV-16/18, overall | 0 | 6
  HPV-16, overall: number analyzed (Participants) | 2167 | 2131
  HPV-16, overall | 0 | 3
  HPV-18, overall: number analyzed (Participants) | 2203 | 2165
  HPV-18, overall | 0 | 4

10. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 and/or -18 Cervical Infection Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN1+ was defined as CIN grades 1, 2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Detection was done in:
  * DNA- and sero-/+: subjects HPV deoxyribonucleic acid (DNA) negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative/positive (sero-/+) for HPV-16 and/or HPV-18 by Enzyme-linked Immunosorbent Assay (ELISA) at baseline (Month 0).
  * Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
Time Frame: Up to Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2224 | 2190
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1898 | 1854
  HPV-16/18, DNA- and sero- subjects | 1 | 7
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1545 | 1521
  HPV-16, DNA- and sero- subjects | 0 | 5
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1597 | 1571
  HPV-18, DNA- and sero- subjects | 1 | 3
  HPV-16/18, DNA- and sero+ subjects: number analyzed (Participants) | 900 | 864
  HPV-16/18, DNA- and sero+ subjects | 0 | 3
  HPV-16, DNA- and sero+ subjects: number analyzed (Participants) | 605 | 594
  HPV-16, DNA- and sero+ subjects | 0 | 1
  HPV-18, DNA- and sero+ subjects: number analyzed (Participants) | 574 | 550
  HPV-18, DNA- and sero+ subjects | 0 | 2
  HPV-16/18, overall | 1 | 11
  HPV-16, overall: number analyzed (Participants) | 2167 | 2131
  HPV-16, overall | 0 | 6
  HPV-18, overall: number analyzed (Participants) | 2203 | 2165
  HPV-18, overall | 1 | 6

11. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 and/or -18 Cervical Infection Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN1+ was defined as CIN grades 1, 2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Detection was done on all subjects irrespective of their baseline HPV DNA and serostatus.
Time Frame: Up to Month 48
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2740 | 2737
Participants
  HPV-16/18 | 35 | 56
  HPV-16 | 24 | 42
  HPV-18 | 13 | 20

12. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Irrespective of HPV Cervical Infection and Irrespective of Baseline HPV DNA Status
Description: CIN1+ was defined as CIN grades 1, 2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Detection was done on all subjects irrespective of their baseline HPV DNA status.
Time Frame: Up to Month 48
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2740 | 2737
Participants | 152 | 178

13. Secondary Outcome: Number of Subjects With Any Cytological Abnormalities Associated With HPV-16 or HPV-18 Cervical Infection
Description: Cytological abnormalities = atypical squamous cells of undetermined significance (ASC-US).
  Detection was done in:
  * DNA- and sero-: subjects HPV deoxyribonucleic acid (DNA) negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative (sero-) for HPV-16 and/or HPV-18 by Enzyme-linked Immunosorbent Assay (ELISA) at baseline (Month 0).
  * Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
  Results for seropositive status were not analysed.
Time Frame: Up to Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2224 | 2190
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1898 | 1854
  HPV-16/18, DNA- and sero- subjects | 2 | 31
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1545 | 1521
  HPV-16, DNA- and sero- subjects | 2 | 24
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1597 | 1571
  HPV-18, DNA- and sero- subjects | 0 | 8
  HPV-16/18, overall | 5 | 38
  HPV-16: number analyzed (Participants) | 2167 | 2131
  HPV-16 | 4 | 27
  HPV-18: number analyzed (Participants) | 2203 | 2165
  HPV-18 | 1 | 12

14. Secondary Outcome: Number of Subjects With Cytological Abnormalities Associated With Oncogenic HPV Types Individually or in Combinations
Description: Oncogenic HPV types included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Detection was done in subjects who were HPV DNA negative for the corresponding HPV type at baseline (at month 0 and Month 6) regardless of initial serostatus.
  HRW-HPV= All high-risk (oncogenic) HPV types excluding HPV-16 and HPV-18 HPV-HR= High-risk (oncogenic) HPV types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68
Time Frame: Up to Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2225 | 2192
Participants
  HPV-16: number analyzed (Participants) | 2167 | 2131
  HPV-16 | 4 | 27
  HPV-18: number analyzed (Participants) | 2203 | 2165
  HPV-18 | 1 | 12
  HPV-31: number analyzed (Participants) | 2172 | 2170
  HPV-31 | 4 | 12
  HPV-33: number analyzed (Participants) | 2204 | 2173
  HPV-33 | 4 | 4
  HPV-35: number analyzed (Participants) | 2211 | 2181
  HPV-35 | 4 | 10
  HPV-39: number analyzed (Participants) | 2196 | 2156
  HPV-39 | 10 | 11
  HPV-45: number analyzed (Participants) | 2206 | 2168
  HPV-45 | 3 | 17
  HPV-51: number analyzed (Participants) | 2171 | 2149
  HPV-51 | 21 | 18
  HPV-52: number analyzed (Participants) | 2158 | 2139
  HPV-52 | 19 | 19
  HPV-56: number analyzed (Participants) | 2200 | 2158
  HPV-56 | 9 | 19
  HPV-58: number analyzed (Participants) | 2198 | 2172
  HPV-58 | 12 | 6
  HPV-59: number analyzed (Participants) | 2202 | 2164
  HPV-59 | 4 | 15
  HPV-66: number analyzed (Participants) | 2187 | 2160
  HPV-66 | 13 | 26
  HPV-68: number analyzed (Participants) | 2184 | 2164
  HPV-68 | 8 | 8
  HPV-31/45: number analyzed (Participants) | 2221 | 2190
  HPV-31/45 | 7 | 28
  HPV-31/45/33/52/58 | 40 | 54
  HPV-39/45/59/68 | 24 | 48
  HPV-31/33/35/52/58 | 41 | 49
  HPV-31/45/33/52/58/35/39/51/56/59 | 79 | 107
  HPV-HRW | 94 | 126
  HPV-HR | 96 | 148

15. Secondary Outcome: Number of Subjects With Histopathologically Confirmed Reduction of Local Cervical Therapy
Description: Detection was done on all subjects irrespective of their baseline HPV DNA status.
Time Frame: Up to Month 48
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2740 | 2737
Participants | 76 | 84

16. Secondary Outcome: Number of Subjects With First Colposcopy
Description: Detection was done on all subjects irrespective of their baseline HPV DNA status.
Time Frame: Up to Month 48
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2741 | 2738
Participants | 392 | 422

17. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Human Papillomavirus (HPV)-16 or HPV-18 and/or With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 and/or -18 Cervical Infection
Description: Persistent cervical HPV infection (6-month definition) was defined as the detection of the same HPV type(s) by polymerase chain reaction (PCR) in cervical samples at 2 consecutive evaluations over approximately a 6-month interval.
  CIN1+ was defined as CIN grades 1, 2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Detection was done on all subjects irrespective of their baseline HPV DNA and serostatus.
Time Frame: Up to Month 48
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2772 | 2779
Participants
  HPV-16/18 | 90 | 158
  HPV-16 | 64 | 118
  HPV-18 | 30 | 52

18. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With HPV-16 or HPV-18 and/or With Histopathologically-confirmed CIN1+ Associated With HPV-16 and/or -18 Cervical Infection Detected Using the HPV Type Assignment Algorithm (TAA).
Description: Persistent cervical HPV infection (6-month definition) was defined as the detection of the same HPV type(s) by polymerase chain reaction (PCR) in cervical samples at 2 consecutive evaluations over approximately a 6-month interval.
  Detection was done on all subjects irrespective of their baseline HPV DNA and serostatus.
  The lesion was assigned to an HPV type found in the lesion if (1) the same HPV type was found in at least 1 of the 2 (closest) preceding cytology samples, or (2) none of the HPV types found in the lesion were found in any of the 2 preceding cytology samples (isolate HPV types)
Time Frame: Up to Month 48
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2772 | 2779
Participants
  HPV-16/18 | 89 | 155
  HPV-16 | 63 | 117
  HPV-18 | 29 | 49

19. Secondary Outcome: Number of Seroconverted Subjects Against HPV-16 in the Immunogenicity Subset.
Description: Seroconversion was defined as the appearance of antibodies (i.e.; titre greater than or equal to the cut-off value) in the serum of subjects seronegative before vaccination.
  HPV-16 assay cut-off value was defined as greater than or equal to 8 ELISA units per millilitre (EL.U/mL). Seronegative (Sero-) subjects are subjects who had an antibody concentration below 8 EL.U/mL prior to vaccination. Seropositive (Sero+) subjects are subjects who had an antibody concentration equal to or above 8 EL.U/mL prior to vaccination.
  Immuno subset=subjects from selected sites N≥1000, at least 250 per region
Time Frame: At pre-vaccination and at Month 7, 12, 18, 24, 36, 48, 60, 72 and 84
Population: The According-To-Protocol cohort for immunogenicity included subjects for whom immunogenicity data were available and for whom assay results were available for antibodies against at least 1 study vaccine antigen component after vaccination. The 15% subset of women enrolled with prior history of HPV disease/infection was included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 406 | 374
Participants
  Sero- before vaccination | 0 | 0
  Sero- at Month 7: number analyzed (Participants) | 406 | 371
  Sero- at Month 7 | 406 | 13
  Sero- at Month 12: number analyzed (Participants) | 384 | 349
  Sero- at Month 12 | 384 | 28
  Sero- at Month 18: number analyzed (Participants) | 377 | 340
  Sero- at Month 18 | 377 | 9
  Sero- at Month 24: number analyzed (Participants) | 392 | 350
  Sero- at Month 24 | 392 | 11
  Sero- at Month 36: number analyzed (Participants) | 361 | 320
  Sero- at Month 36 | 361 | 23
  Sero- at Month 48: number analyzed (Participants) | 345 | 316
  Sero- at Month 48 | 345 | 31
  Sero- at Month 60: number analyzed (Participants) | 275 | 251
  Sero- at Month 60 | 275 | 11
  Sero- at Month 72: number analyzed (Participants) | 277 | 260
  Sero- at Month 72 | 276 | 5
  Sero- at Month 84: number analyzed (Participants) | 275 | 255
  Sero- at Month 84 | 273 | 2
  Sero+ before vaccination: number analyzed (Participants) | 170 | 179
  Sero+ before vaccination | 170 | 179
  Sero+ at Month 7: number analyzed (Participants) | 170 | 179
  Sero+ at Month 7 | 170 | 166
  Sero+ at Month 12: number analyzed (Participants) | 154 | 158
  Sero+ at Month 12 | 154 | 151
  Sero+ at Month 24: number analyzed (Participants) | 158 | 165
  Sero+ at Month 24 | 158 | 144
  Sero+ at Month 18: number analyzed (Participants) | 147 | 154
  Sero+ at Month 18 | 147 | 136
  Sero+ at Month 36: number analyzed (Participants) | 137 | 146
  Sero+ at Month 36 | 137 | 131
  Sero+ at Month 48: number analyzed (Participants) | 132 | 145
  Sero+ at Month 48 | 132 | 135
  Sero+ at Month 60: number analyzed (Participants) | 99 | 95
  Sero+ at Month 60 | 99 | 79
  Sero+ at Month 72: number analyzed (Participants) | 99 | 102
  Sero+ at Month 72 | 99 | 57
  Sero+ at Month 84: number analyzed (Participants) | 95 | 101
  Sero+ at Month 84 | 95 | 51

20. Secondary Outcome: Number of Seroconverted Subjects Against HPV-18 in the Immunogenicity Subset.
Description: Seroconversion was defined as the appearance of antibodies (i.e.; titre greater than or equal to the cut-off value) in the serum of subjects seronegative before vaccination.
  HPV-18 assay cut-off value was defined as greater than or equal to 7 ELISA units per millilitre (EL.U/mL). Seronegative (Sero-) subjects are subjects who had an antibody concentration below 7 EL.U/mL prior to vaccination. Seropositive (Sero+) subjects are subjects who had an antibody concentration equal to or above 7 EL.U/mL prior to vaccination.
  Immuno subset=subjects from selected sites N≥1000, at least 250 per region
Time Frame: At pre-vaccination and at Month 7, 12, 18, 24, 36, 48, 60, 72 and 84
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 405 | 379
Participants
  Sero- before vaccination | 0 | 0
  Sero- at Month 7: number analyzed (Participants) | 405 | 374
  Sero- at Month 7 | 405 | 12
  Sero- at Month 12: number analyzed (Participants) | 376 | 352
  Sero- at Month 12 | 375 | 16
  Sero- at Month 18: number analyzed (Participants) | 366 | 347
  Sero- at Month 18 | 366 | 12
  Sero- at Month 24: number analyzed (Participants) | 389 | 358
  Sero- at Month 24 | 387 | 14
  Sero- at Month 36: number analyzed (Participants) | 348 | 328
  Sero- at Month 36 | 346 | 14
  Sero- at Month 48: number analyzed (Participants) | 338 | 320
  Sero- at Month 48 | 336 | 16
  Sero- at Month 60: number analyzed (Participants) | 268 | 246
  Sero- at Month 60 | 266 | 11
  Sero- at Month 72: number analyzed (Participants) | 269 | 254
  Sero- at Month 72 | 261 | 3
  Sero- at month 84: number analyzed (Participants) | 268 | 248
  Sero- at month 84 | 257 | 3
  Sero+ before vaccination: number analyzed (Participants) | 163 | 164
  Sero+ before vaccination | 163 | 164
  Sero+ at Month 7: number analyzed (Participants) | 163 | 161
  Sero+ at Month 7 | 163 | 146
  Sero+ at Month 12: number analyzed (Participants) | 154 | 144
  Sero+ at Month 12 | 154 | 133
  Sero+ at Month 18: number analyzed (Participants) | 149 | 141
  Sero+ at Month 18 | 149 | 118
  Sero+ at Month 24: number analyzed (Participants) | 153 | 150
  Sero+ at Month 24 | 153 | 114
  Sero+ at Month 36: number analyzed (Participants) | 142 | 131
  Sero+ at Month 36 | 142 | 92
  Sero+ at Month 48: number analyzed (Participants) | 133 | 131
  Sero+ at Month 48 | 133 | 94
  Sero+ at Month 60: number analyzed (Participants) | 101 | 91
  Sero+ at Month 60 | 101 | 58
  Sero+ at Month 72: number analyzed (Participants) | 103 | 99
  Sero+ at Month 72 | 103 | 32
  Sero+ at Month 84: number analyzed (Participants) | 98 | 98
  Sero+ at Month 84 | 98 | 32

21. Secondary Outcome: Geometric Mean Concentrations (GMCs) Against HPV-16 Antibody in the Immunogenicity Subset.
Description: GMCs were expressed in ELISA units per milliliter (EL.U/mL).
  Seronegative (Sero-) subjects are subjects who had an antibody concentration below 8 EL.U/mL prior to vaccination. Seropositive (Sero+) subjects are subjects who had an antibody concentration equal to or above 8 EL.U/mL prior to vaccination.
  Immuno subset=subjects from selected sites (N≥1000, at least 250 per region)
Time Frame: At pre-vaccination and at Month 7, 12, 18, 24, 36, 48, 60, 72 and 84
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 406 | 374
EL.U/mL
  Sero-before vaccination | NA [NA to NA] — Not calculable as no subject had HPV-16 antibody concentration equal to or above the assay cut-off value. | NA [NA to NA] — Not calculable as no subject had HPV-16 antibody concentration equal to or above the assay cut-off value.
  Sero- at Month 7: number analyzed (Participants) | 406 | 371
  Sero- at Month 7 | 5412.9 [4934.3 to 5938.0] | 4.3 [4.1 to 4.4]
  Sero- at Month 12: number analyzed (Participants) | 384 | 349
  Sero- at Month 12 | 1542.5 [1393.2 to 1707.8] | 4.4 [4.2 to 4.5]
  Sero- at Month 18: number analyzed (Participants) | 377 | 340
  Sero- at Month 18 | 992.6 [893.9 to 1102.2] | 4.1 [4.0 to 4.2]
  Sero- at Month 24: number analyzed (Participants) | 392 | 350
  Sero- at Month 24 | 827.8 [745.2 to 919.5] | 4.2 [4.1 to 4.4]
  Sero- at Month 36: number analyzed (Participants) | 361 | 320
  Sero- at Month 36 | 612.9 [550.1 to 682.8] | 4.5 [4.2 to 4.7]
  Sero- at Month 48: number analyzed (Participants) | 345 | 316
  Sero- at Month 48 | 546.2 [490.4 to 608.2] | 4.6 [4.4 to 4.9]
  Sero- at Month 60: number analyzed (Participants) | 275 | 251
  Sero- at Month 60 | 447.1 [394.3 to 507.0] | 4.3 [4.1 to 4.5]
  Sero- at Month 72: number analyzed (Participants) | 277 | 260
  Sero- at Month 72 | 412.8 [364.0 to 468.1] | 9.8 [9.5 to 10.0]
  Sero- at Month 84: number analyzed (Participants) | 275 | 255
  Sero- at Month 84 | 381.0 [334.7 to 433.8] | 9.6 [9.4 to 9.9]
  Sero+ before vaccination: number analyzed (Participants) | 170 | 179
  Sero+ before vaccination | 39.3 [33.6 to 45.9] | 38.6 [33.2 to 44.9]
  Sero+ at Month 7: number analyzed (Participants) | 170 | 179
  Sero+ at Month 7 | 5845.5 [5113.8 to 6682.0] | 33.4 [28.2 to 39.5]
  Sero+ at month 12: number analyzed (Participants) | 154 | 158
  Sero+ at month 12 | 2705.8 [2313.2 to 3165.1] | 38.0 [32.0 to 45.3]
  Sero+ at Month 18: number analyzed (Participants) | 147 | 154
  Sero+ at Month 18 | 2104.7 [1780.5 to 2487.8] | 30.5 [25.2 to 36.9]
  Sero+ at Month 24: number analyzed (Participants) | 158 | 165
  Sero+ at Month 24 | 1883.5 [1599.4 to 2218.1] | 29.6 [24.5 to 35.7]
  Sero+ at month 36: number analyzed (Participants) | 137 | 146
  Sero+ at month 36 | 1363.8 [1138.2 to 1634.2] | 30.6 [25.3 to 37.0]
  Sero+ at Month 48: number analyzed (Participants) | 132 | 145
  Sero+ at Month 48 | 1261.2 [1048.4 to 1517.1] | 34.3 [28.8 to 40.8]
  Sero+ at Month 60: number analyzed (Participants) | 99 | 95
  Sero+ at Month 60 | 943.0 [749.2 to 1187.0] | 24.7 [19.2 to 31.7]
  Sero+ at Month 72: number analyzed (Participants) | 99 | 102
  Sero+ at Month 72 | 1053.7 [841.0 to 1320.3] | 25.6 [20.7 to 31.5]
  Sero+ at Month 84: number analyzed (Participants) | 95 | 101
  Sero+ at Month 84 | 954.3 [755.3 to 1205.8] | 23.9 [19.3 to 29.5]

22. Secondary Outcome: Geometric Mean Concentrations (GMCs) Against HPV-18 Antibody in the Immunogenicity Subset.
Description: GMCs were expressed in ELISA units per milliliter (EL.U/mL).
  Seronegative (Sero-) subjects are subjects who had an antibody concentration below 7 EL.U/mL prior to vaccination. Seropositive (Sero+) subjects are subjects who had an antibody concentration equal to or above 7 EL.U/mL prior to vaccination.
  Immuno subset=subjects from selected sites (N≥1000, at least 250 per region)
Time Frame: At pre-vaccination and at Month 7, 12, 18, 24, 36, 48, 60, 72 and 84
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 405 | 379
EL.U/mL
  Sero- before vaccination | NA [NA to NA] — Not calculable as no subject had HPV-18 antibody concentration equal to or above the assay cut-off value. | NA [NA to NA] — Not calculable as no subject had HPV-18 antibody concentration equal to or above the assay cut-off value.
  Sero- at Month 7: number analyzed (Participants) | 405 | 374
  Sero- at Month 7 | 2567.7 [2339.5 to 2818.2] | 3.7 [3.6 to 3.9]
  Sero- at Month 12: number analyzed (Participants) | 376 | 352
  Sero- at Month 12 | 645.3 [576.6 to 722.1] | 3.7 [3.6 to 3.9]
  Sero- at Month 18: number analyzed (Participants) | 366 | 347
  Sero- at Month 18 | 402.6 [359.7 to 450.6] | 3.7 [3.6 to 3.8]
  Sero- at Month 24: number analyzed (Participants) | 389 | 358
  Sero- at Month 24 | 321.7 [286.9 to 360.7] | 3.7 [3.6 to 3.9]
  Sero- at Month 36: number analyzed (Participants) | 348 | 328
  Sero- at Month 36 | 245.9 [218.5 to 276.8] | 3.7 [3.6 to 3.8]
  Sero- at Month 48: number analyzed (Participants) | 338 | 320
  Sero- at Month 48 | 228.5 [201.9 to 258.7] | 3.7 [3.6 to 3.8]
  Sero- at Month 60: number analyzed (Participants) | 268 | 246
  Sero- at Month 60 | 174.3 [151.2 to 200.8] | 3.8 [3.6 to 4.0]
  Sero- at Month 72: number analyzed (Participants) | 269 | 254
  Sero- at Month 72 | 177.7 [154.1 to 204.8] | 9.2 [9.0 to 9.5]
  Sero- at Month 84: number analyzed (Participants) | 268 | 248
  Sero- at Month 84 | 166.2 [143.4 to 192.7] | 9.1 [9.0 to 9.3]
  Sero+ before vaccination: number analyzed (Participants) | 163 | 164
  Sero+ before vaccination | 23.0 [19.9 to 26.7] | 24.2 [20.6 to 28.4]
  Sero+ at Month 7: number analyzed (Participants) | 163 | 161
  Sero+ at Month 7 | 2933.9 [2557.1 to 3366.3] | 21.9 [18.1 to 26.5]
  Sero+ at Month 12: number analyzed (Participants) | 154 | 144
  Sero+ at Month 12 | 936.2 [796.4 to 1100.4] | 23.6 [19.4 to 28.7]
  Sero+ at Month 18: number analyzed (Participants) | 149 | 141
  Sero+ at Month 18 | 661.3 [560.9 to 779.7] | 19.5 [15.7 to 24.2]
  Sero+ at Month 24: number analyzed (Participants) | 153 | 150
  Sero+ at Month 24 | 573.6 [487.7 to 674.6] | 16.6 [13.5 to 20.5]
  Sero+ at Month 36: number analyzed (Participants) | 142 | 131
  Sero+ at Month 36 | 423.1 [357.9 to 500.1] | 16.4 [12.9 to 20.7]
  Sero+ at Month 48: number analyzed (Participants) | 133 | 131
  Sero+ at Month 48 | 392.3 [328.9 to 468.0] | 15.9 [12.7 to 19.9]
  Sero+ at Month 60: number analyzed (Participants) | 101 | 91
  Sero+ at Month 60 | 306.0 [245.7 to 380.9] | 12.9 [9.8 to 16.9]
  Sero+ at Month 72: number analyzed (Participants) | 103 | 99
  Sero+ at Month 72 | 324.8 [264.3 to 399.1] | 16.2 [13.3 to 19.6]
  Sero+ at Month 84: number analyzed (Participants) | 98 | 98
  Sero+ at Month 84 | 302.2 [243.4 to 375.2] | 16.5 [13.4 to 20.4]

23. Secondary Outcome: Number of Seroconverted Subjects Against HPV-16 and HPV-18 Viral Neutralization in a Selected Subset of Subjects.
Description: Seroconversion was defined as the appearance of antibodies (i.e.; titre greater than or equal to the cut-off value) in the serum of subjects seronegative before vaccination. HPV-16/18 assay cut-off value was defined as greater than or equal to 40 Estimated dose 50% (ED50). Sero- subjects are subjects who had an antibody concentration below 40 ED50 prior to vaccination. Sero+ subjects are subjects who had an antibody concentration equal to or above 50 ED50 prior to vaccination. ED50 = the estimated serum dilution reducing the signal generated by viral infection by 50%
Time Frame: Prior to vaccination and at Months 7, 12, 18, 24, 48 and 84.
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 38 | 37
Participants
  HPV-16 sero- [pre-vaccination]: number analyzed (Participants) | 37 | 37
  HPV-16 sero- [pre-vaccination] | 0 | 0
  HPV-16 sero- [at Month 7]: number analyzed (Participants) | 37 | 37
  HPV-16 sero- [at Month 7] | 37 | 1
  HPV-16 sero- [at Month 12]: number analyzed (Participants) | 37 | 37
  HPV-16 sero- [at Month 12] | 37 | 0
  HPV-16 sero- [at Month 18]: number analyzed (Participants) | 36 | 37
  HPV-16 sero- [at Month 18] | 36 | 0
  HPV-16 sero- [at Month 24]: number analyzed (Participants) | 35 | 37
  HPV-16 sero- [at Month 24] | 35 | 2
  HPV-16 sero- [at Month 48]: number analyzed (Participants) | 27 | 33
  HPV-16 sero- [at Month 48] | 27 | 1
  HPV-16 sero- [at Month 84]: number analyzed (Participants) | 20 | 25
  HPV-16 sero- [at Month 84] | 19 | 1
  HPV-16 sero+ [pre-vaccination]: number analyzed (Participants) | 4 | 1
  HPV-16 sero+ [pre-vaccination] | 4 | 1
  HPV-16 sero+ [at Month 7]: number analyzed (Participants) | 4 | 1
  HPV-16 sero+ [at Month 7] | 4 | 1
  HPV-16 sero+ [at Month 12]: number analyzed (Participants) | 4 | 1
  HPV-16 sero+ [at Month 12] | 4 | 1
  HPV-16 sero+ [at Month 18]: number analyzed (Participants) | 4 | 1
  HPV-16 sero+ [at Month 18] | 4 | 1
  HPV-16 sero+ [at Month 24]: number analyzed (Participants) | 4 | 1
  HPV-16 sero+ [at Month 24] | 4 | 0
  HPV-16 sero+ [at Month 48]: number analyzed (Participants) | 3 | 1
  HPV-16 sero+ [at Month 48] | 3 | 0
  HPV-16 sero+ [at Month 84]: number analyzed (Participants) | 3 | 1
  HPV-16 sero+ [at Month 84] | 3 | 1
  HPV-18 sero- [pre-vaccination]: number analyzed (Participants) | 38 | 35
  HPV-18 sero- [pre-vaccination] | 0 | 0
  HPV-18 sero- [at Month 7]: number analyzed (Participants) | 38 | 35
  HPV-18 sero- [at Month 7] | 38 | 0
  HPV-18 sero- [at Month 12]: number analyzed (Participants) | 38 | 35
  HPV-18 sero- [at Month 12] | 38 | 0
  HPV-18 sero- [at Month 18]: number analyzed (Participants) | 37 | 35
  HPV-18 sero- [at Month 18] | 37 | 0
  HPV-18 sero- [at Month 24]: number analyzed (Participants) | 36 | 35
  HPV-18 sero- [at Month 24] | 36 | 1
  HPV-18 sero- [at Month 48]: number analyzed (Participants) | 29 | 32
  HPV-18 sero- [at Month 48] | 29 | 0
  HPV-18 sero- [at Month 84]: number analyzed (Participants) | 22 | 25
  HPV-18 sero- [at Month 84] | 22 | 0
  HPV-18 sero+ [pre-vaccination]: number analyzed (Participants) | 3 | 3
  HPV-18 sero+ [pre-vaccination] | 3 | 3
  HPV-18 sero+ [at Month 7]: number analyzed (Participants) | 3 | 3
  HPV-18 sero+ [at Month 7] | 3 | 2
  HPV-18 sero+ [at Month 12]: number analyzed (Participants) | 3 | 3
  HPV-18 sero+ [at Month 12] | 3 | 2
  HPV-18 sero+ [at Month 18]: number analyzed (Participants) | 3 | 3
  HPV-18 sero+ [at Month 18] | 3 | 2
  HPV-18 sero+ [at Month 24]: number analyzed (Participants) | 3 | 3
  HPV-18 sero+ [at Month 24] | 3 | 2
  HPV-18 sero+ [at Month 48]: number analyzed (Participants) | 1 | 2
  HPV-18 sero+ [at Month 48] | 1 | 1
  HPV-18 sero+ [at Month 84]: number analyzed (Participants) | 1 | 1
  HPV-18 sero+ [at Month 84] | 1 | 1

24. Secondary Outcome: Geometric Mean Titers (GMTs) Against HPV-16 and HPV-18 Viral Neutralization Antibodies in a Selected Subset of Subjects.
Description: Titers are expressed as geometric mean antibody titers (GMTs).
  Seronegative (Sero-) subjects are subjects who had an antibody titer below 40 ED50 prior to vaccination. Seropositive (Sero+) subjects are subjects who had an antibody titer equal to or above 40 ED50 prior to vaccination.
  ED50 = Estimated dose 50%, the estimated serum dilution reducing the signal generated by viral infection by 50%
Time Frame: Prior to vaccination and at Months 7, 12, 18, 24, 48 and 84.
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 38 | 37
Titers
  HPV-16 sero- [pre-vaccination] | NA [NA to NA] — Not calculable as no subject had HPV-16 antibody titer equal to or above the assay cut-off value. | NA [NA to NA] — Not calculable as no subject had HPV-16 antibody titer equal to or above the assay cut-off value.
  HPV-16 sero- [at Month 7]: number analyzed (Participants) | 37 | 37
  HPV-16 sero- [at Month 7] | 11663.5 [7507.2 to 18120.8] | 20.8 [19.2 to 22.4]
  HPV-16 sero- [at Month 12]: number analyzed (Participants) | 37 | 37
  HPV-16 sero- [at Month 12] | 5597.7 [3688.3 to 8495.6] | NA [NA to NA] — Not calculable as no subject had HPV-16 antibody titer equal to or above the assay cut-off value.
  HPV-16 sero- [at Month 18]: number analyzed (Participants) | 36 | 37
  HPV-16 sero- [at Month 18] | 2175.2 [1390.8 to 3401.9] | NA [NA to NA] — Not calculable as no subject had HPV-16 antibody titer equal to or above the assay cut-off value.
  HPV-16 sero- [at Month 24]: number analyzed (Participants) | 35 | 37
  HPV-16 sero- [at Month 24] | 1941.7 [1193.0 to 3160.4] | 22.3 [18.6 to 26.6]
  HPV-16 sero- [at Month 48]: number analyzed (Participants) | 27 | 33
  HPV-16 sero- [at Month 48] | 828.9 [488.4 to 1406.7] | 21.4 [18.7 to 24.5]
  HPV-16 sero- [at Month 84]: number analyzed (Participants) | 20 | 37
  HPV-16 sero- [at Month 84] | 1213.4 [1213.4 to 2779.1] | NA [NA to NA] — Not calculable as no subject had HPV-16 antibody titer equal to or above the assay cut-off value.
  HPV-16 sero+ [pre-vaccination]: number analyzed (Participants) | 4 | 37
  HPV-16 sero+ [pre-vaccination] | 139.3 [32.7 to 594.2] | 45.0 [NA to NA] — Data were not calculable because of too few subjects.
  HPV-16 sero+ [at Month 7]: number analyzed (Participants) | 4 | 37
  HPV-16 sero+ [at Month 7] | 20283.2 [2428.3 to 169422.0] | 107.0 [NA to NA] — Data were not calculable because of too few subjects.
  HPV-16 sero+ [at Month 12]: number analyzed (Participants) | 4 | 37
  HPV-16 sero+ [at Month 12] | 19484.3 [7049.3 to 53854.2] | 99.0 [NA to NA] — Data were not calculable because of too few subjects.
  HPV-16 sero+ [at Month 18]: number analyzed (Participants) | 4 | 37
  HPV-16 sero+ [at Month 18] | 4393.3 [798.4 to 24175.0] | 93.0 [NA to NA] — Data were not calculable because of too few subjects.
  HPV-16 sero+ [at Month 24]: number analyzed (Participants) | 4 | 37
  HPV-16 sero+ [at Month 24] | 9459.1 [2168.4 to 41263.7] | NA [NA to NA] — Not calculable as no subject had HPV-16 antibody titer equal to or above the assay cut-off value.
  HPV-16 sero+ [at Month 48]: number analyzed (Participants) | 3 | 37
  HPV-16 sero+ [at Month 48] | 4187.2 [676.4 to 25921.6] | NA [NA to NA] — Not calculable as no subject had HPV-16 antibody titer equal to or above the assay cut-off value.
  HPV-16 sero+ [at Month 84]: number analyzed (Participants) | 3 | 37
  HPV-16 sero+ [at Month 84] | 5837.0 [5837.0 to 35354.6] | NA [NA to NA] — Not calculable as no subject had HPV-16 antibody titer equal to or above the assay cut-off value.
  HPV-18 sero- [pre-vaccination] | NA [NA to NA] — Not calculable as no subject had HPV-18 antibody titer equal to or above the assay cut-off value. | NA [NA to NA] — Not calculable as no subject had HPV-18 antibody titer equal to or above the assay cut-off value.
  HPV-18 sero- [at Month 7] | 7959.6 [4648.0 to 13630.7] | NA [NA to NA] — Not calculable as no subject had HPV-18 antibody titer equal to or above the assay cut-off value.
  HPV-18 sero- [at Month 12] | 1979.9 [1201.6 to 3262.5] | NA [NA to NA] — Not calculable as no subject had HPV-18 antibody titer equal to or above the assay cut-off value.
  HPV-18 sero- [at Month 18]: number analyzed (Participants) | 37 | 37
  HPV-18 sero- [at Month 18] | 1334.6 [793.3 to 2245.3] | NA [NA to NA] — Not calculable as no subject had HPV-18 antibody titer equal to or above the assay cut-off value.
  HPV-18 sero- [at Month 24]: number analyzed (Participants) | 36 | 35
  HPV-18 sero- [at Month 24] | 826.6 [493.6 to 1384.1] | 21.4 [18.7 to 24.5]
  HPV-18 sero- [at Month 48]: number analyzed (Participants) | 29 | 37
  HPV-18 sero- [at Month 48] | 386.1 [203.9 to 731.1] | NA [NA to NA] — Not calculable as no subject had HPV-18 antibody titer equal to or above the assay cut-off value.
  HPV-18 sero- [at Month 84]: number analyzed (Participants) | 22 | 37
  HPV-18 sero- [at Month 84] | 491.2 [232.9 to 1036.0] | NA [NA to NA] — Not calculable as no subject had HPV-18 antibody titer equal to or above the assay cut-off value.
  HPV-18 sero+ [pre-vaccination]: number analyzed (Participants) | 3 | 3
  HPV-18 sero+ [pre-vaccination] | 84.7 [9.2 to 782.4] | 115.5 [21.5 to 621.0]
  HPV-18 sero+ [at Month 7]: number analyzed (Participants) | 3 | 3
  HPV-18 sero+ [at Month 7] | 3014.5 [446.3 to 20361.5] | 163.4 [0.8 to 31959.2]
  HPV-18 sero+ [at Month 12]: number analyzed (Participants) | 3 | 3
  HPV-18 sero+ [at Month 12] | 3377.8 [2563.9 to 4450.1] | 167.3 [0.8 to 35164.4]
  HPV-18 sero+ [at Month 18]: number analyzed (Participants) | 3 | 3
  HPV-18 sero+ [at Month 18] | 3125.8 [595.8 to 16398.4] | 254.9 [0.4 to 172814.0]
  HPV-18 sero+ [at Month 24]: number analyzed (Participants) | 3 | 3
  HPV-18 sero+ [at Month 24] | 2493.0 [261.2 to 23793.7] | 154.9 [0.4 to 53341.9]
  HPV-18 sero+ [at Month 48]: number analyzed (Participants) | 38 | 2
  HPV-18 sero+ [at Month 48] | 545.0 [NA to NA] — Data were not calculable because of too few subjects. | 86.0 [0.0 to 9662500000]
  HPV-18 sero+ [at Month 84] | NA [NA to NA] — Data were not calculable because of too few subjects. | 968.0 [NA to NA] — Data were not calculable because of too few subjects.

25. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as pain that prevented normal activity. Grade 3 redness and swelling was defined as redness/swelling above 50 millimeter (mm).
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented and symptom sheets completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2830 | 2831
Participants
  Any pain | 2411 | 1862
  Grade 3 pain | 303 | 73
  Any redness | 1058 | 530
  Grade 3 redness | 44 | 5
  Any swelling | 1080 | 428
  Grade 3 swelling | 97 | 11

26. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal, headache, myalgia, rash, urticaria and fever (Fever = axillary temperature above 37.5 degrees Celsius (°C)). Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 urticaria = urticaria distributed on at least 4 body areas. Grade 3 fever = axillary temperature above 39.0°C.
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2832 | 2832
Participants
  Any arthralgia | 580 | 439
  Grade3 arthralgia | 30 | 24
  Related arthralgia | 323 | 225
  Any fatigue | 1116 | 916
  Grade 3 fatigue | 78 | 53
  Related fatigue | 678 | 545
  Any fever | 308 | 248
  Grade 3 fever | 17 | 8
  Related fever | 181 | 159
  Any gastrointestinal | 664 | 592
  Grade 3 gastrointestinal | 60 | 54
  Related gastrointestinal | 335 | 312
  Any headache | 1165 | 1074
  Grade 3 headache | 76 | 72
  Related headache | 666 | 598
  Any myalgia | 878 | 622
  Grade 3 myalgia | 46 | 32
  Related myalgia | 541 | 391
  Any rash | 185 | 124
  Grade 3 rash | 1 | 7
  Related rash | 88 | 61
  Any urticaria | 258 | 201
  Grade 3 urticaria | 21 | 18
  Related urticaria | 84 | 79

27. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Grade 3 unsolicited AE = an event that prevented normal activity.
  A related AE = event assessed by the investigator as causally related to the study vaccination.
Time Frame: Within 30 days (Days 0 - 29) post-vaccination period.
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2877 | 2870
Participants
  Any AEs | 1153 | 1164
  Grade 3 AEs | 208 | 184
  Related AEs | 246 | 191

28. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects. A related SAE was defined as an event assessed by the investigator as causally related to the study vaccination.
Time Frame: Up to Month 48 and up to Month 84
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2877 | 2870
Participants
  Any SAEs, M48 | 286 | 266
  Related SAEs, M48 | 5 | 8
  Any SAEs, M84 | 291 | 269
  Related SAEs, M84 | 5 | 8

29. Secondary Outcome: Number of Subjects Reporting Related or Fatal Serious Adverse Event.
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Up to Month 84
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2877 | 2870
Participants
  Fatal AEs | 13 | 5
  Related SAEs | 5 | 8

30. Secondary Outcome: Number of Subjects Reporting Any AE/SAE Leading to Premature Discontinuation of the Study.
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
  Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Up to Month 84
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2877 | 2870
Participants | 28 | 14

31. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Disease (NOCDs).
Description: NOCDs include autoimmune disorders, asthma and type I diabetes.
Time Frame: Up to Month 48
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2877 | 2870
Participants | 143 | 165

32. Secondary Outcome: Number of Subjects Reporting New Onset of Autoimmune Disease (NOADs).
Time Frame: Up to Month 48
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2877 | 2870
Participants | 24 | 24

33. Secondary Outcome: Number of Subjects Reporting Medically Significant Conditions (MAEs).
Description: Medically significant conditions were defined as: AEs prompting emergency room or physician visits that were not (1) related to common diseases or (2) routine visits for physical examination or vaccination, or SAEs that were not related to common diseases. Common diseases included: upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervicovaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: Up to Month 48
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2877 | 2870
Participants | 1170 | 1140

34. Secondary Outcome: Number of Subjects With Pregnancies and Their Outcomes.
Description: Pregnancy outcomes are live infant, premature live infant, elective termination, ectopic pregnancy, spontaneous abortion, lost to follow-up and pregnancy ongoing. For each category it was specified if the infant presents congenital anomaly (CA) or no apparent congenital anomaly (No ACA).
Time Frame: Up to Month 48
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 359 | 357
Participants
  Live infant No ACA, M48 | 259 | 249
  Live infant CA, M48 | 4 | 7
  Elective termination No ACA, M48 | 19 | 24
  Elective termination CA, M48 | 1 | 0
  Ectopic pregnancy, M48 | 5 | 6
  Spontaneous abortion No ACA, M48 | 69 | 66
  Spontaneous abortion CA, M48 | 0 | 1
  Stillbirth No ACA, M48 | 0 | 2
  Lost to follow-up, M48 | 2 | 2

35. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 and/or -18 Cervical Infection Detected Using the Type Assignment Algorithm (TAA)
Description: CIN1+ was defined as CIN grades 1, 2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Detection was done on subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
  TAA: Type assignment algorithm. The lesion was assigned to an HPV type found in the lesion if
  1. the same HPV type was found in at least one of the two (closest) preceding cytology samples, or
  2. none of the HPV types found in the lesion were found in any of the two preceding cytology samples (isolate HPV types)
Time Frame: Up to Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2224 | 2190
Participants
  HPV-16/18 DNA- | 1 | 9
  HPV-16 DNA-: number analyzed (Participants) | 2167 | 2131
  HPV-16 DNA- | 0 | 5
  HPV-18 DNA-: number analyzed (Participants) | 2203 | 2165
  HPV-18 DNA- | 1 | 5

36. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Human Papillomavirus (HPV)-16 or HPV-18
Description: Persistent cervical HPV infection (6-month definition) was defined as the detection of the same HPV type(s) by PCR in cervical samples at 2 consecutive evaluations over approximately a 6-month interval. Detection was done in: - DNA- and sero-/+: subjects HPV DNA negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative/positive (sero-/+) for HPV-16 and/or HPV-18 by ELISA at baseline (Month 0). - Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
Time Frame: Up to Month 84
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2124 | 2109
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1815 | 1786
  HPV-16/18, DNA- and sero- subjects | 6 | 67
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1482 | 1466
  HPV-16, DNA- and sero- subjects | 5 | 51
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1535 | 1511
  HPV-18, DNA- and sero- subjects | 1 | 17
  HPV-16/18, DNA- and sero+ subjects: number analyzed (Participants) | 851 | 837
  HPV-16/18, DNA- and sero+ subjects | 3 | 13
  HPV-16, DNA- and sero+ subjects: number analyzed (Participants) | 574 | 573
  HPV-16, DNA- and sero+ subjects | 2 | 9
  HPV-18, DNA- and sero+ subjects: number analyzed (Participants) | 541 | 534
  HPV-18, DNA- and sero+ subjects | 1 | 4
  HPV-16/18, overall | 9 | 82
  HPV-16, overall: number analyzed (Participants) | 2073 | 2055
  HPV-16, overall | 7 | 60
  HPV-18, overall: number analyzed (Participants) | 2108 | 2085
  HPV-18, overall | 2 | 23

37. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With Human Papillomavirus (HPV)-16 or HPV-18
Description: Persistent cervical HPV infection (12-month definition) was defined as the detection of the same HPV type(s) PCR in cervical samples at all available time points over approximately a 12-month interval (evaluations are planned at approximately 6-month intervals). - DNA- and sero-/+: subjects HPV DNA negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative/positive (sero-/+) for HPV-16 and/or HPV-18 by ELISA at baseline (Month 0). - Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
Time Frame: Up to Month 84
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2093 | 2081
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1789 | 1764
  HPV-16/18, DNA- and sero- subjects | 2 | 37
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1464 | 1447
  HPV-16, DNA- and sero- subjects | 1 | 27
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1513 | 1494
  HPV-18, DNA- and sero- subjects | 1 | 10
  HPV-16/18, DNA- and sero+ subjects: number analyzed (Participants) | 835 | 825
  HPV-16/18, DNA- and sero+ subjects | 0 | 5
  HPV-16, DNA- and sero+ subjects: number analyzed (Participants) | 562 | 567
  HPV-16, DNA- and sero+ subjects | 0 | 3
  HPV-18, DNA- and sero+ subjects: number analyzed (Participants) | 532 | 523
  HPV-18, DNA- and sero+ subjects | 0 | 2
  HPV-16/18, overall | 2 | 43
  HPV-16, overall: number analyzed (Participants) | 2043 | 2030
  HPV-16, overall | 1 | 30
  HPV-18, overall: number analyzed (Participants) | 2077 | 2057
  HPV-18, overall | 1 | 13

38. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Oncogenic HPV Types Individually or in Combinations.
Description: as for outcome 7
Time Frame: Up to Month 84
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2125 | 2111
Participants
  HPV-16: number analyzed (Participants) | 2073 | 2055
  HPV-16 | 7 | 60
  HPV-18: number analyzed (Participants) | 2108 | 2085
  HPV-18 | 2 | 23
  HPV-31: number analyzed (Participants) | 2073 | 2090
  HPV-31 | 10 | 29
  HPV-33: number analyzed (Participants) | 2105 | 2094
  HPV-33 | 12 | 9
  HPV-35: number analyzed (Participants) | 2112 | 2101
  HPV-35 | 11 | 17
  HPV-39: number analyzed (Participants) | 2097 | 2078
  HPV-39 | 34 | 26
  HPV-45: number analyzed (Participants) | 2106 | 2088
  HPV-45 | 9 | 30
  HPV-51: number analyzed (Participants) | 2071 | 2072
  HPV-51 | 48 | 42
  HPV-52: number analyzed (Participants) | 2060 | 2058
  HPV-52 | 54 | 56
  HPV-56: number analyzed (Participants) | 2100 | 2081
  HPV-56 | 28 | 30
  HPV-58: number analyzed (Participants) | 2098 | 2092
  HPV-58 | 24 | 19
  HPV-59: number analyzed (Participants) | 2105 | 2083
  HPV-59 | 22 | 21
  HPV-66: number analyzed (Participants) | 2089 | 2080
  HPV-66 | 45 | 49
  HPV-68: number analyzed (Participants) | 2084 | 2085
  HPV-68 | 31 | 33
  HPV-31/45: number analyzed (Participants) | 2121 | 2109
  HPV-31/45 | 19 | 57
  HPV-31/45/33/52/58 | 98 | 128
  HPV-39/45/59/68 | 92 | 102
  HPV-31/33/35/52/58 | 101 | 118
  HPV-31/45/33/52/58/35/39/51/56/59 | 206 | 220
  HPV-HRW | 255 | 274
  HPV-HR | 262 | 330

39. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With Oncogenic HPV Types Individually or in Combinations.
Description: Oncogenic HPV types included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68. subjects HPV DNA- for the corresponding HPV type at Month 0 6, regardless of initial serostatus. HPV-HRW=All high-risk (oncogenic) HPV types excluding HPV-16 and HPV-18 HPV-HR=High-risk (oncogenic) HPV types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 , 68
Time Frame: Up to Month 84
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2094 | 2083
Participants
  HPV-16: number analyzed (Participants) | 2043 | 2030
  HPV-16 | 1 | 30
  HPV-18: number analyzed (Participants) | 2077 | 2057
  HPV-18 | 1 | 13
  HPV-31: number analyzed (Participants) | 2044 | 2062
  HPV-31 | 7 | 17
  HPV-33: number analyzed (Participants) | 2074 | 2068
  HPV-33 | 9 | 7
  HPV-35: number analyzed (Participants) | 2081 | 2073
  HPV-35 | 5 | 9
  HPV-39: number analyzed (Participants) | 2067 | 2050
  HPV-39 | 20 | 10
  HPV-45: number analyzed (Participants) | 2076 | 2060
  HPV-45 | 7 | 13
  HPV-51: number analyzed (Participants) | 2040 | 2045
  HPV-51 | 23 | 26
  HPV-52: number analyzed (Participants) | 2029 | 2031
  HPV-52 | 34 | 31
  HPV-56: number analyzed (Participants) | 2071 | 2054
  HPV-56 | 11 | 15
  HPV-58: number analyzed (Participants) | 2067 | 2065
  HPV-58 | 14 | 13
  HPV-59: number analyzed (Participants) | 2074 | 2055
  HPV-59 | 7 | 10
  HPV-66: number analyzed (Participants) | 2058 | 2052
  HPV-66 | 22 | 16
  HPV-68: number analyzed (Participants) | 2053 | 2057
  HPV-68 | 13 | 22
  HPV-31/45: number analyzed (Participants) | 2091 | 2081
  HPV-31/45 | 14 | 28
  HPV-31/45/33/52/58 | 65 | 75
  HPV-39/45/59/68 | 46 | 54
  HPV-31/33/35/52/58 | 64 | 72
  HPV-31/45/33/52/58/35/39/51/56/59 | 118 | 129
  HPV-HRW | 145 | 160
  HPV-HR | 147 | 194

40. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)2+ Associated With HPV-16 and/or -18 Cervical Infection Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN2+ was defined as CIN grades 2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer. Detection was done in: - DNA- and sero-: subjects HPV deoxyribonucleic acid (DNA) negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative (sero-) for HPV-16 and/or HPV-18 by Enzyme-linked Immunosorbent Assay (ELISA) at baseline (Month 0). - Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline. Note: Results for seropositive status were not analysed.
Time Frame: Up to Month 84
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2168 | 2146
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1852 | 1818
  HPV-16/18, DNA- and sero- subjects | 1 | 6
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1507 | 1491
  HPV-16, DNA- and sero- subjects | 1 | 5
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1565 | 1541
  HPV-18, DNA- and sero- subjects | 1 | 2
  HPV-16/18, overall | 1 | 8
  HPV-16, overall: number analyzed (Participants) | 2112 | 2090
  HPV-16, overall | 1 | 5
  HPV-18, overall: number analyzed (Participants) | 2149 | 2122
  HPV-18, overall | 1 | 4

41. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 and/or -18 Cervical Infection Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN1+ was defined as CIN grades 1, 2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer. Detection was done in: - DNA- and sero-/+: subjects HPV deoxyribonucleic acid (DNA) negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative/positive (sero-/+) for HPV-16 and/or HPV-18 by Enzyme-linked Immunosorbent Assay (ELISA) at baseline (Month 0). - Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
Time Frame: Up to Month 84
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2168 | 2146
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1852 | 1818
  HPV-16/18, DNA- and sero- subjects | 2 | 12
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1507 | 1491
  HPV-16, DNA- and sero- subjects | 1 | 9
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1565 | 1541
  HPV-18, DNA- and sero- subjects | 2 | 4
  HPV-16/18, DNA- and sero+ subjects: number analyzed (Participants) | 870 | 848
  HPV-16/18, DNA- and sero+ subjects | 0 | 3
  HPV-16, DNA- and sero+ subjects: number analyzed (Participants) | 588 | 583
  HPV-16, DNA- and sero+ subjects | 0 | 1
  HPV-18, DNA- and sero+ subjects: number analyzed (Participants) | 552 | 539
  HPV-18, DNA- and sero+ subjects | 0 | 2
  HPV-16/18, overall | 2 | 16
  HPV-16, overall: number analyzed (Participants) | 2112 | 2090
  HPV-16, overall | 1 | 10
  HPV-18, overall: number analyzed (Participants) | 2149 | 2122
  HPV-18, overall | 2 | 7

42. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 and/or -18 Cervical Infection Detected Within the Lesional Component of the Cervical Tissue Specimen
Time Frame: Up to Month 84
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2733 | 2735
Participants
  HPV-16/18 | 37 | 66
  HPV-16 | 26 | 49
  HPV-18 | 14 | 23

43. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Irrespective of HPV Cervical Infection and Irrespective of Baseline HPV DNA Status
Description: as for outcome 12
Time Frame: Up to Month 84
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2733 | 2735
Participants | 179 | 229

44. Secondary Outcome: Number of Subjects With Any Cytological Abnormalities Associated With HPV-16 or HPV-18 Cervical Infection
Description: Cytological abnormalities = atypical squamous cells of undetermined significance (ASC-US). Detection was done in: - DNA- and sero-: subjects HPV deoxyribonucleic acid (DNA) negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative (sero-) for HPV-16 and/or HPV-18 by Enzyme-linked Immunosorbent Assay (ELISA) at baseline (Month 0). - Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline. Results for seropositive status were not analysed.
Time Frame: Up to Month 84
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2168 | 2146
Participants
  HPV-16/18, DNA- and sero- subjects: number analyzed (Participants) | 1852 | 1818
  HPV-16/18, DNA- and sero- subjects | 3 | 47
  HPV-16, DNA- and sero- subjects: number analyzed (Participants) | 1507 | 1491
  HPV-16, DNA- and sero- subjects | 3 | 34
  HPV-18, DNA- and sero- subjects: number analyzed (Participants) | 1565 | 1541
  HPV-18, DNA- and sero- subjects | 0 | 14
  HPV-16/18, overall | 6 | 56
  HPV-16: number analyzed (Participants) | 2112 | 2090
  HPV-16 | 5 | 38
  HPV-18: number analyzed (Participants) | 2149 | 2122
  HPV-18 | 1 | 19

45. Secondary Outcome: Number of Subjects With Cytological Abnormalities Associated With Oncogenic HPV Types Individually or in Combinations
Description: as for outcome 14
Time Frame: Up to Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2169 | 2148
Participants
  HPV-16: number analyzed (Participants) | 2112 | 2090
  HPV-16 | 5 | 38
  HPV-18: number analyzed (Participants) | 2149 | 2122
  HPV-18 | 1 | 19
  HPV-31: number analyzed (Participants) | 2117 | 2127
  HPV-31 | 5 | 23
  HPV-33: number analyzed (Participants) | 2149 | 2130
  HPV-33 | 6 | 8
  HPV-35: number analyzed (Participants) | 2156 | 2137
  HPV-35 | 7 | 13
  HPV-39: number analyzed (Participants) | 2141 | 2114
  HPV-39 | 21 | 23
  HPV-45: number analyzed (Participants) | 2150 | 2125
  HPV-45 | 5 | 23
  HPV-51: number analyzed (Participants) | 2115 | 2107
  HPV-51 | 38 | 34
  HPV-52: number analyzed (Participants) | 2103 | 2095
  HPV-52 | 25 | 22
  HPV-56: number analyzed (Participants) | 2114 | 2115
  HPV-56 | 15 | 28
  HPV-58: number analyzed (Participants) | 2142 | 2128
  HPV-58 | 19 | 13
  HPV-59: number analyzed (Participants) | 2147 | 2120
  HPV-59 | 9 | 22
  HPV-66: number analyzed (Participants) | 2133 | 2117
  HPV-66 | 22 | 43
  HPV-68: number analyzed (Participants) | 2128 | 2120
  HPV-68 | 15 | 15
  HPV-31/45: number analyzed (Participants) | 2165 | 2146
  HPV-31/45 | 10 | 44
  HPV-31/45/33/52/58 | 56 | 78
  HPV-39/45/59/68 | 49 | 74
  HPV-31/33/35/52/58 | 56 | 70
  HPV-31/45/33/52/58/35/39/51/56/59 | 119 | 160
  HPV-HRW | 143 | 192
  HPV-HR | 145 | 223

46. Secondary Outcome: Number of Subjects With Histopathologically Confirmed Reduction of Local Cervical Therapy
Description: Detection was done on all subjects irrespective of their baseline HPV DNA status.
Time Frame: Up to Month 84
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Groups:
- Aluminium Hydroxide: Subjects received 3 doses of Aluminium Hydroxide [Al(OH)3]. Aluminium Hydroxide was administered intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6 months schedule.
Arm/Group | Cervarix Group | Aluminium Hydroxide
Number analyzed (Participants) | 2733 | 2735
Participants | 88 | 110

47. Secondary Outcome: Number of Subjects With First Colposcopy
Description: Detection was done on all subjects irrespective of their baseline HPV DNA status.
Time Frame: Up to Month 84
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2734 | 2736
Participants | 506 | 560

48. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Human Papillomavirus (HPV)-16 or HPV-18 and/or With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 and/or -18 Cervical Infection
Description: as for outcome 17
Time Frame: Up to Month 84
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2768 | 2778
Participants
  HPV-16/18 | 93 | 209
  HPV-16 | 66 | 152
  HPV-18 | 32 | 71

49. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With HPV-16 or HPV-18 and/or With Histopathologically-confirmed CIN1+ Associated With HPV-16 and/or -18 Cervical Infection Detected Using the HPV Type Assignment Algorithm (TAA).
Description: as for outcome 18
Time Frame: Up to Month 84
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Number analyzed (Participants) | 2768 | 2778
Participants
  HPV-16/18 | 92 | 206
  HPV-16 | 65 | 151
  HPV-18 | 30 | 68

ADVERSE EVENTS:
Time Frame: SAEs: from the beginning of the study up to Month 84. Unsolicited AEs: within 30 days (Days 0-29) post-vaccination period). Solicited AEs: During the 7-day (Days 0-6) post-vaccination period.
Arm/Group | Cervarix Group | Aluminium Hydroxide Group
Serious Adverse Events (participants affected / at risk) | 291/2881 | 269/2871
Other Adverse Events (participants affected / at risk) | 2543/2881 | 2236/2871
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=2881) | Aluminium Hydroxide Group (N=2871)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 19 | 16
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 19 | 13
Appendicitis (Infections and infestations) | 13 | 12
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 13 | 12
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 9
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 10 | 11
Cholelithiasis (Hepatobiliary disorders) | 5 | 9
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 6 | 7
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 4 | 7
Ovarian cyst (Reproductive system and breast disorders) | 5 | 6
Dengue fever (Infections and infestations) | 9 | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 7 | 2
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 5
Gastroenteritis (Infections and infestations) | 5 | 3
Urinary tract infection (Infections and infestations) | 5 | 3
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Pyelonephritis (Infections and infestations) | 6 | 1
Hypertension (Vascular disorders) | 4 | 2
Suicide attempt (Psychiatric disorders) | 5 | 1
Uterine polyp (Reproductive system and breast disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Cholecystitis (Hepatobiliary disorders) | 3 | 2
Nephrolithiasis (Renal and urinary disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 3
Menorrhagia (Reproductive system and breast disorders) | 1 | 4
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 3
Premature labour (Pregnancy, puerperium and perinatal conditions) | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pyelonephritis acute (Infections and infestations) | 3 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 2
Depression (Psychiatric disorders) | 2 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 2
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 3
Endometriosis (Reproductive system and breast disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 2 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pneumonia (Infections and infestations) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 1
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Diarrhoea infectious (Gastrointestinal disorders) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Goitre (Endocrine disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Salpingitis (Infections and infestations) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Migraine (Nervous system disorders) | 5 | 0
Convulsion (Nervous system disorders) | 0 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Cholecystitis acute (Hepatobiliary disorders) | 3 | 0
Completed suicide (Psychiatric disorders) | 3 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 3
Anaphylactic reaction (Immune system disorders) | 0 | 2
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 2
Bronchopneumonia (Infections and infestations) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Major depression (Psychiatric disorders) | 0 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 2
Ovarian cyst torsion (Reproductive system and breast disorders) | 2 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Sinusitis (Infections and infestations) | 2 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Addison's disease (Endocrine disorders) | 0 | 1
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Adnexal torsion (Reproductive system and breast disorders) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amniotic cavity infection (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Anaesthetic complication pulmonary (Injury, poisoning and procedural complications) | 1 | 0
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 1
Anorexia nervosa (Psychiatric disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Bartholinitis (Reproductive system and breast disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 1
Basedow's disease (Endocrine disorders) | 1 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchogenic cyst (Congenital, familial and genetic disorders) | 0 | 1
Burn infection (Infections and infestations) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cerebral cyst (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chest pain (General disorders) | 1 | 0
Chlamydial infection (Infections and infestations) | 0 | 1
Cholesterosis (Metabolism and nutrition disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Immune system disorders) | 0 | 1
Colpocele (Reproductive system and breast disorders) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Conversion disorder (Psychiatric disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Cystitis klebsiella (Infections and infestations) | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1
Diabetic coma (Nervous system disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Endosalpingiosis (Reproductive system and breast disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Epiploic appendagitis (Gastrointestinal disorders) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Genital prolapse (Reproductive system and breast disorders) | 1 | 0
Genitourinary tract infection (Infections and infestations) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Homicide (Social circumstances) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Ill-defined disorder (General disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Incarcerated hernia (General disorders) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Intracranial haematoma (Nervous system disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Lyme disease (Infections and infestations) | 1 | 0
Macular oedema (Eye disorders) | 1 | 0
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 1
Opisthorchiasis (Infections and infestations) | 0 | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pasteurella infection (Infections and infestations) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Placenta accreta (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Placental transfusion syndrome (Blood and lymphatic system disorders) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 1
Polymyalgia rheumatica (Reproductive system and breast disorders) | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1
Pyonephrosis (Infections and infestations) | 0 | 1
Pyrexia (Gastrointestinal disorders) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Renal abscess (Infections and infestations) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Retinal vein thrombosis (Eye disorders) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1
Sedation (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Thyroid cyst (Endocrine disorders) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Typhoid fever (Infections and infestations) | 1 | 0
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0
Uterine atony (Reproductive system and breast disorders) | 0 | 1
Uterine cyst (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Vertebral artery dissection (Nervous system disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 2
Viral infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=2881) | Aluminium Hydroxide Group (N=2871)
Headache (Nervous system disorders) | 203 | 222
Pain (General disorders) | 2411 | 1862
Redness (General disorders) | 1058 | 530
Swelling (General disorders) | 1080 | 428
Arthralgia (General disorders) | 580 | 439
Fatigue (General disorders) | 1116 | 916
Fever (General disorders) | 308 | 248
Gastrointestinal (General disorders) | 664 | 592
Headache (General disorders) | 1165 | 1074
Myalgia (General disorders) | 878 | 622
Rash (General disorders) | 185 | 124
Urticaria (General disorders) | 258 | 201

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.